CLINICAL TRIAL: NCT00884962
Title: A Dose Ranging Study of the Aeris Polymeric Lung Volume Reduction (PLVR) System in Patients With Advanced Upper Lobe Predominant Emphysema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-C08-003PLV
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Advanced Emphysema
Keywords: emphysema; aeris; PLVR; BLVR; germany; treatment; device; breathing
MeSH Terms: conditions — Emphysema; Respiratory Aspiration

ARMS (1):
- PLVR (Experimental)
  Interventions: Device: Polymeric Lung Volume Reduction System (PLVR)

INTERVENTIONS:
Device: Polymeric Lung Volume Reduction System (PLVR) — 20ml (each) of polymer will be injected into 2, 3 or 4 subsegments during the first treatment. Eligible patients may have 20ml (each) of polymer will be injected into 2 or 3 subsegments during the second treatment.

SUMMARY:
This is a multi-center, open-label, non-controlled Pilot Study. Approximately 24 patients will be assigned to one of 3 treatment groups (8 patients each group). Patients in each group will receive 2, 4, and 6 (3 followed by a retreatment of 3) subsegmental treatments, respectively. All patients will receive treatment in a single lung under conscious sedation or general anesthesia. Patients will be followed for 24 weeks after completion of PLVR treatment(s). Upon completion of 12-week follow-up, all safety and efficacy data will be analyzed to determine an effective treatment dose. Thereafter, Group 1 patients may elect to be retreated at additional sites so that their total dose received is consistent with the effective dose. All study patients will receive standard medical therapy in addition to PLVR.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of advanced upper lobe predominant (ULP) emphysema or advanced disease in the superior lower lobes as defined by FEV1/FVC <70 % predicted, FEV1 of < 50% predicted, TLC > 100% of predicted, and RV > 135% predicted.
* Patients must have persistent symptoms despite medical therapy and either not be candidates for Lung Volume Reduction Surgery (LVRS) or have elected not to undergo LVRS.
* Patients must be > 40 years of age, have symptoms despite medical therapy, and have none of the pre-specified co-morbid conditions that could influence study outcomes or their ability to tolerate bronchoscopy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in the ratio of Residual Volume (RV) to Total Lung Capacity (TLC) | 12 and 24 weeks following treatment
  Change from baseline in RV/TLC ratio at 12 and 24 weeks following treatment

SECONDARY OUTCOMES:
Change in Forced Expiratory Volume in 1 Second (FEV1) | 12 and 24 weeks following treatment
  o Change from baseline in FEV1 (post bronchodilator) at 12 and 24 weeks following treatment
Change in Forced Vital Capacity (FVC) | 12 and 24 weeks following treatment
  Change from baseline in FVC (post bronchodilator) at 12 and 24 weeks following treatment
Change in Diffusing Capacity of the Lung for Carbon Monoxide (DLco) | 12 and 24 weeks following treatment
  Change from baseline in DLco at 12 and 24 weeks following treatment
Change in Medical Research Council Dyspnea (MRCD) score | 12 and 24 weeks following treatment
  Change from baseline in MRCD score at 12 and 24 weeks
Change in distance walked in six minutes | 12 and 24 weeks following treatment
  Change from baseline at 12 and 248 weeks in 6 Minutes Walk Test (6MWT)
Change in St. George's Respiratory Questionnaire (SGRQ) domain score | 12 and 24 weeks following treatment
  Change from baseline in disease-specific health related quality of life assessment (SGRQ) at 12 and 24 weeks following treatment

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Chefarzt Klinik für Pneumologie, Bad Berka
  - Charité Universitätsmedizin Medizinische Klinik Infektiologie und Pulmologie, Berlin
  - Pneumologisches Forschungsinstitut, Großhansdorf
  - Thoraxklinik Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Medizinische Klinik und Poliklinik Klinikum Großhadern, Munich

REFERENCES:
- [Derived] Agrawal A. Interventional Pulmonology: Diagnostic and Therapeutic Advances in Bronchoscopy. Am J Ther. 2021 Feb 9;28(2):e204-e216. doi: 10.1097/MJT.0000000000001344. PMID 33590989
- [Derived] Magnussen H, Kramer MR, Kirsten AM, Marquette C, Valipour A, Stanzel F, Bonnet R, Behr J, Fruchter O, Refaely Y, Eberhardt R, Herth FJ. Effect of fissure integrity on lung volume reduction using a polymer sealant in advanced emphysema. Thorax. 2012 Apr;67(4):302-8. doi: 10.1136/thoraxjnl-2011-201038. Epub 2012 Feb 28. PMID 22374920